CLINICAL TRIAL: NCT01210781
Title: Target Planning for Placement of DBS-electrodes and Follow-up of the Clinical Efficacy of Stimulation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: DBS
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Movement Disorders; Epilepsy
Keywords: All indication for deep brain stimulation (DBS)
MeSH Terms: conditions — Movement Disorders; Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: deep brain stimulation (DBS) — deep brain stimulation (DBS) is in itself not part of this study but a clinical indication. The study aims at documenting DBS parameters and outcome

SUMMARY:
Deep brain stimulation (DBS) has been established as therapy for severe forms of Parkinson's disease and other indications. A common target for stimulation is the subthalamic nucleus (STN). Nevertheless, there is no agreement on the mechanisms how DBS leads to clinical improvement.

The project aims to describe the variability of target coordinates in the patient group and to relate it to clinical outcome as documented in standardized questionaires.

* Trial with surgical intervention

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) has been established as therapy for severe forms of Parkinson's disease and other indications. A common target for stimulation is the subthalamic nucleus (STN). Nevertheless, there is no agreement on the mechanisms how DBS leads to clinical improvement.

The project aims to describe the variability of target coordinates in the patient group and to relate it to clinical outcome as documented in standardized questionaires.

ELIGIBILITY:
Inclusion criteria:

* Patients fullfill all criteria for implantation of deep brain stimulation (DBS) electrodes
* Patients are able to give informed written consent

Exclusion criteria:

* Patients do not their give informed written consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients implanted with DBS electrodes at our institution
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
neurological outcome | 5 years
  UPDRS

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sarnthein, Prof Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery
Locations (1):
- University Hospital Zurich, Neurosurgery, Zurich, Canton of Zurich, Switzerland